CLINICAL TRIAL: NCT00501488
Title: Effect of Adiponectin Genetic Polymorphism on Rosiglitazone Response
Status: Completed | Type: Observational
Sponsor: Central South University (Other)
Other Study IDs: Zhao-Qian Liu
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2007-07-20 (Estimated); Status verified 2007-07

CONDITIONS: Diabetes Mellitus
Keywords: pharmacodynamics; insulin resistance; therapy; volunteer
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Rosiglitazone

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: rosiglitazone

SUMMARY:
The aims of the present study were to investigate the association between adiponectin gene polymorphisms and the response to rosiglitazone monotherapy in T2D patients.

A total of 255 T2D patients and 120 health volunteers were enrolled in this study. 42 T2D patients with -11377(C/G) or +45(T/G) genotypes were selected to administrate orally 4mg rosiglitazone daily for 12 consecutive weeks.

DETAILED DESCRIPTION:
The aims of the present study were to investigate the association between adiponectin allele +45(T/G) and -11377(C/G) polymorphisms and the response to rosiglitazone monotherapy in T2D patients.

A total of 255 T2D patients (138 males, 117 females) aged from 25 to 70 years (mean 48.6 ± 10.7 years) and 120 healthy controls (53 females, 67 males) aged from 25 to 70 years(mean 47.1 ± 11.0 years) were enrolled to participate in this study. Physical examination, medical history and serum biochemical tests were performed to identify healthy or T2D subjects. The diagnosis criteria of T2D patients were made according to the World Health Organization in 1997 by fasting plasma glucose (FPG  7.0 mmol/L) and/or postprandial plasma glucose test (PPG  11.1 mmol/L). The inclusion criteria of all subjects were that subjects had the range of body mass index (BMI) from 18.5 to 30 kg/m2 and did not administrate any PPAR agonists in the last 3 months. Patients who were receiving insulin treatment, pregnant or lactating women, or with serious diseases such as acute myocardial infarction, cerebral vascular accident, trauma, and kidney disease or liver disease were excluded from this study. Table 1 showed the characteristic profiles of T2D patients and healthy controls. There were no statistical differences in the age, height, weight, and BMI value between T2D patients and healthy controls. All subjects were recruited from local residents in Changsha city, Hunan Province, P. R. China. The study protocol was approved by the Ethics Committee of Xiangya School of Medicine, Central South University and written informed consents were obtained before the start of this study. A total of 42 T2D patients (23 male, 19 female) were randomly selected to be only treated with 4mg rosiglitazone daily for 12 consecutive weeks without change in previous medications.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis criteria of T2D patients were made according to the World Health Organization in 1997 by fasting plasma glucose (FPG  7.0 mmol/L) and/or postprandial plasma glucose test (PPG  11.1 mmol/L)
* The inclusion criteria of all subjects were that subjects had the range of body mass index (BMI) from 18.5 to 30 kg/square meter and did not administrate any PPAR agonists in the last 3 months.

Exclusion Criteria:

* Patients who were receiving insulin treatment, pregnant or lactating women, or with serious diseases such as acute myocardial infarction, cerebral vascular accident, trauma, and kidney disease or liver disease were excluded from this study.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-03; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhao-Qian Liu, MD, Ph.D, Principal Investigator — Central South University Xiangya School of Medicine
Locations (1):
- Central South University, Changsha, Hunan, China

REFERENCES:
- See also: Related Info — http://www.csupharmacol.com